CLINICAL TRIAL: NCT06912646
Title: An Evaluation of the Effect of the Erchonia® EVRL™ for Prescription Home Use Application in Providing Temporary Relief From Idiopathic Peripheral Neuropathy Foot Pain
Brief Title: Clinical Efficacy of the Erchonia EVRL for Providing Temporary Relief of Idiopathic Peripheral Neuropathy Foot Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-IPN
Record Dates: First submitted 2025-04-03; First posted 2025-04-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Neuropathy; Neuropathy;Peripheral
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Erchonia® EVRL™ (Experimental): The Erchonia® EVRL™ is made up of (1) 635 nanometers red laser diode and (1) 405 nanometers violet laser diode mounted in a portable handheld device.
  Interventions: Device: Erchonia® EVRL™

INTERVENTIONS:
Device: Erchonia® EVRL™ — The Erchonia® EVRL™ is made up of (1) 635 nanometers red laser diode and (1) 405 nanometers violet laser diode mounted in a portable handheld device. The diodes are positioned approximately 3 to 6 inches from the top of the foot. The treatments will be self-administered by the subject at his or her's place of residence, two times per day for 21 days. Each procedure administration lasts 5 minutes per foot, for a total of 10 minutes.

SUMMARY:
The purpose of this clinical study is to determine the effectiveness of the Erchonia® EVRL™, manufactured by Erchonia Corporation (the Company), in providing prescription home use application for temporary relief of idiopathic neuropathy foot pain in individuals diagnosed with idiopathic neuropathy by a suitably qualified and licensed health professional.

DETAILED DESCRIPTION:
This clinical study is a single-arm, active treatment group only, non-inferiority prospective design to evaluate the efficacy of the Erchonia® EVRL™ for prescription home use application in providing temporary relief of foot pain due to idiopathic peripheral neuropathy. There will be a single active treatment only subject group in this study. All enrolled subjects will self-administer the treatments with the active (true) Erchonia® EVRL™ laser in his or her own home.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with idiopathic peripheral neuropathy by a suitably qualified and licensed health professional within the past 6 months.
* Over the age of 22 years of age
* Able to read and write English
* Constant feet pain on-going over at least the past 3 months
* Subjects using analgesics (pain medication) must be on a stable analgesic regimen (i.e., no changes to the prescribed analgesic regimen) over a period of at least 14 days prior to study enrollment; and be willing and able to not have planned upward dose titration of analgesics during the study period. Decreasing frequency of analgesic use during the study is permitted. Cannabis prescribed for medicinal purposes qualifies as an analgesic in this context
* Willing and able to refrain from engaging in any non-study therapies for the management of foot pain throughout the course of study participation, including conventional therapies such as physical therapy, occupational therapy, hot or cold packs, and alternative therapies such as chiropractic care and acupuncture
* Agrees to refrain from taking a dosage of analgesic (pain medication) for at least 6 hours before a scheduled VAS foot pain rating is to be recorded
* Subject's degree of foot pain on the 0-100 VAS, with "0" being no pain and "100" being worst pain imaginable, is 50 or greater

Exclusion Criteria:

* Diabetic, referred to as having hemoglobin A1c (HbA1C) of 6.5% or higher
* Previously diagnosed with any definitive (i.e. not idiopathic) cause of peripheral neuropathy by a suitably qualified and licensed health professional within the past 6 months, such as diabetes, injury, infection, toxins and poisons, alcoholism, medications such as chemotherapy, autoimmune disorders, etc..
* Pregnant or possibly pregnant, breastfeeding, or planning pregnancy during the intended course of study participation
* Open wounds (sores, cuts, ulcers, etc.) on or around the treatment area on the feet
* Cancerous growths or lesions on or around the treatment area on the feet
* Difficulty with hand dexterity sufficient to negatively impact the ability to administer treatments with the laser such as from severe arthritis in the hands, Multiple Sclerosis, Cerebral Palsy, Parkinson's Disease, Huntington's Disease, etc.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-16 (Estimated); Study Completion 2027-06-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With a 30% or Greater Change in Pain Rating on the Visual Analog Scale | Baseline and 3 weeks
  The Visual Analog Scale (VAS) will be used to assess pain from baseline to the 6-week endpoint for each subject. Subjects will be instructed to indicate the overall level of pain experienced in their feet by placing a cross (X) on a 10-centimeter horizontal line. The left end of the line will be labeled "0," representing "no pain," and the right end will be labeled "100," representing "the worst pain imaginable." Individual subject success is defined as a 30% or greater change in VAS pain scores across the evaluation period. A negative (-) percent change indicates a decrease in pain level and is positive for individual subject success. A lower VAS pain score from baseline to study endpoint represents a better outcome, whereas a higher score from baseline to study endpoint represents a worse outcome.

SECONDARY OUTCOMES:
Neuropathic Pain Symptom Inventory | Baseline and 3 weeks
  The Neuropathic Pain Symptom Inventory (NPSI) is a 12-item self-administered patient-reported outcome assessment tool with a recall/ observation period of over the past 24 hours. It contains 10 descriptors representing 5 distinct dimensions on the basis of factor analysis: burning pain, deep pain, paroxysmal pain, evoked pain, paresthesia/dysesthesia, and 2 temporal items designed to assess pain duration and the number of pain paroxysms. The NPSI has a maximum total score of 100, a lower score from baseline to study endpoint represents a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Franco & Co, Miramar, Florida, United States

IPD SHARING:
Plan to Share IPD: No